CLINICAL TRIAL: NCT07143630
Title: Effects of Abdominal Electrical Stimulation on Balance and Ultrasound-Measured Muscle Thickness in Stroke Patients: A Prospective Randomized Controlled Trials
Brief Title: Abdominal Electrical Stimulation for Balance and Muscle Thickness in Stroke Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Başakşehir Çam & Sakura City Hospital (Other Government)
Responsible Party: Principal Investigator, tuba sarıkaya, Resident in Physical Medicine and Rehabilitation, Başakşehir Çam & Sakura City Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 26.02.2025.79
Record Dates: First submitted 2025-08-20; First posted 2025-08-27 (Actual); Last update posted 2025-09-03 (Actual); Status verified 2025-08

CONDITIONS: Stroke
Keywords: postural balance; balance impairment; rehabilitation; neuromuscular electrical stimulation; abdominal muscle
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Intervention Model Description: This study is a prospective, randomized, parallel-group trial. Stroke patients will be randomly assigned to one of two groups: (1) an intervention group receiving neuromuscular electrical stimulation (NMES) applied to the abdominal muscles in addition to core stabilization exercises, or (2) a control group performing only core stabilization exercises.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- NMES + Core Stabilization Exercises (Experimental)
  Interventions: Device: Neuromuscular Electrical Stimulation; Behavioral: Core Stabilization Exercises
- Core Stabilization Exercises Only (Active Comparator)
  Interventions: Behavioral: Core Stabilization Exercises

INTERVENTIONS:
Device: Neuromuscular Electrical Stimulation — NMES will be applied to the abdominal muscles using a multichannel stimulator. Each session will last approximately 20 minutes, administered 5 times per week for a total of 15 sessions, in addition to core stabilization exercise program performed with the same frequency.
  Other Names: Chattanooga multichanel stimulator
  Arms: NMES + Core Stabilization Exercises
Behavioral: Core Stabilization Exercises — Participants will perform a structured core stabilization exercise program. The program will be administered 5 times per week for a total of 15 sessions.
  Other Names: Trunk stabilization training

SUMMARY:
Stroke is a leading cause of balance impairment and trunk muscle weakness, which restricts independence in daily activities. Neuromuscular electrical stimulation (NMES) is a safe rehabilitation method to activate muscles. This study will evaluate the effects of NMES applied to the abdominal muscles on balance and ultrasound-measured muscle thickness in stroke patients. The findings may provide evidence for new treatment strategies to enhance trunk function and improve quality of life after stroke.

DETAILED DESCRIPTION:
Stroke is a leading cause of long-term disability and frequently results in impaired balance and trunk muscle weakness, limiting independence in daily life. Abdominal muscles are essential for postural stability, and their weakness may adversely affect mobility and functional outcomes in stroke patients. Neuromuscular electrical stimulation (NMES) is a safe rehabilitation method used to promote muscle contraction and improve strength. While NMES has shown positive effects on limb muscles, its impact on abdominal muscles and balance remains insufficiently studied.

In this prospective randomized controlled trial, participants will be randomly allocated into two groups. The control group will perform core stabilization exercises, while the intervention group will receive core stabilization exercises combined with abdominal NMES. Balance will be assessed using validated clinical scales, and abdominal muscle thickness will be measured by ultrasound. The study aims to determine the additional effects of abdominal NMES on balance, trunk control, and functional recovery in stroke patients.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 65 years.
* At least 1 month since the onset of stroke.
* Ability to maintain sitting balance without support.
* Ability to stand with or without support.
* Voluntary agreement to participate in the study (signed informed consent).

Exclusion Criteria:

* History of hemiplegia on the contralateral side of the body.
* Medically unstable condition.
* History of orthopedic or neurological disease that may cause balance impairment.
* Presence of balance problems prior to stroke.
* Body mass index (BMI) ≥ 35
* Presence of a cardiac pacemaker.
* Diagnosis of malignancy.
* Epilepsy.
* Pregnancy.
* Open wound or infection in the area where stimulation will be applied.
* Lack of cooperation or inability to follow instructions.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Estimated)
Dates: Start 2025-04-01 (Actual); Primary Completion 2025-10-01 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
Change in Balance Performance (Berg Balance Scale) | Baseline and after 15 sessions (≈3 weeks)
  Balance will be assessed using the Berg Balance Scale (BBS; maximum score: 56, minimum score: 0). Higher scores indicate better balance, lower scores indicate worse balance.
Abdominal Muscle Thickness (Ultrasound) | Baseline and after 15 sessions (≈3 weeks)]
  Abdominal muscle thickness will be measured in millimeters by ultrasound at rest. Higher values indicate greater muscle thickness.

SECONDARY OUTCOMES:
Trunk Control (Trunk Control test) | Baseline and after 15 sessions (≈3 weeks)]
Fear of Falling (Visual Analog Scale - VAS) | Baseline and after 15 sessions (≈3 weeks)]
  Fear of falling will be evaluated using a Visual Analog Scale (VAS; score range: 0-10 cm, where 0 = no fear and 10 = maximum fear). Higher scores indicate greater fear of falling.
Change in Postural Control (Postural Assessment Scale for Stroke Patients) | Baseline and after 15 sessions (≈3 weeks)]
  Postural control will be assessed using the Postural Assessment Scale for Stroke Patients (PASS; score range: 0-36). Higher scores indicate better postural control, lower scores indicate worse control.
Functional Ambulation (Functional Ambulation Classification - FAC) | Baseline and after 15 sessions (≈3 weeks)]
  Ambulation will be measured using the Functional Ambulation Classification (FAC; score range: 0-5). Higher scores indicate better functional ambulation.
Mobility (Timed Up and Go Test - TUG) | Baseline and after 15 sessions (≈3 weeks)]
  Mobility will be assessed using the Timed Up and Go Test (TUG; measured in seconds). Lower times indicate better mobility, higher times indicate worse mobility.
Motor Recovery (Brunnstrom Stages) | Baseline and after 15 sessions (≈3 weeks)]
  Motor recovery will be assessed using Brunnstrom Stages of Motor Recovery (score range: Stage 1-6). Higher stages indicate better motor recovery.

CONTACTS AND LOCATIONS:
Overall Officials: Tuba SARIKAYA, Principal Investigator — Başakşehir Çam & Sakura City Hospital
Locations (1):
- Başakşehir Çam and Sakura City Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No